CLINICAL TRIAL: NCT04496466
Title: Clinical Characterization Protocol for Severe Infectious Diseases (CCPSEI)
Acronym: CCPSEI
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00245545
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — As part of a secondary objective, we plan to develop a data and specimen repository that acts as a resource for the investigation and analysis of downstream research questions specific to the clinical course of COVID-19, the development of medical countermeasures and diagnostic tests, and, basic biology questions associated with SARS-CoV-2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a standardized protocol for the rapid, coordinated clinical investigation of severe or potentially severe acute infections by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Participants with acute illness suspected to be caused by SARS-CoV-2 (COVID-19) will be enrolled. This protocol has been designed to enable data and biological samples to be prospectively collected and shared rapidly in a globally-harmonized sampling schedule. Multiple independent studies can be easily aggregated, tabulated and analyzed across many different settings globally. The protocol is the product of many years of discussion among international investigators from a wide range of scientific and medical. Recruitment under this protocol has been initiated in response to Middle Eastern Respiratory Syndrome coronavirus (MERS-CoV) in 2012-2013, Influenza H7N9 in 2013, viral hemorrhagic fever (Ebolavirus) in 2014, Monkeypox & MERS-coronavirus in 2018, Tick-borne encephalitis virus (TBEV) in 2019 and COVID-19 in 2020. Participants may be newly identified through healthcare system or public health access, under quarantine, or in isolation care in outpatient or inpatient settings relevant to the Johns Hopkins University School of Medicine. Other locations may adopt this study concurrently, under a deferred review, or cooperatively.

The existence of this protocol would ensure a timely, comprehensive epidemiologic and clinical characterization of the initial cases of COVID-19 in a mounting pandemic. The World Health Organization (WHO) recognized the need for standardized data collection for the epidemiology, immunology and clinical characteristics of these novel pathogens, and established the International Severe Acute Respiratory and Emerging Infection Consortium (ISARIC) network in 2011. At the core of the protocol are a standardized schedule, structure and content of clinical, laboratory and microbiologic data collection, supplemented by domain-specific components (e.g., acute respiratory infection, viral hemorrhagic fever). The timepoints of this protocol will also be aligned with a separate multi-center institutional review board (IRB) approved protocol to describe patients with emerging infectious diseases that present to military treatment facilities within the United States.

DETAILED DESCRIPTION:
Infectious disease is the single biggest cause of death worldwide. New infectious agents, such as the SARS, MERS and SARS CoV-2, novel influenza viruses, viruses causing viral hemorrhagic fever (e.g. Ebola), and viruses that affect the central nervous system (CNS) such as TBEV & Nipah require investigation to understand pathogen biology and pathogenesis in the host. Even for known infections, resistance to antimicrobial therapies is widespread, and treatments to control potentially deleterious host responses are lacking.

In order to develop a mechanistic understanding of disease processes, such that risk factors for severe illness can be identified and treatments can be developed, it is necessary to understand pathogen characteristics associated with virulence, the replication dynamics and in-host evolution of the pathogen, the dynamics of the host response, the pharmacology of antimicrobial or host-directed therapies, the transmission dynamics, and factors underlying individual susceptibility.

The novel severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has led to almost 500,000 cases of COVID-19 and over 22,000 deaths worldwide. There have been 24,738 cases and 291 deaths in the United states and 190 cases in Maryland, USA as of March 21, 2020. The global is dire, with reports of severe overcrowding in hospitals, shortages of medical supplies, and insufficient medical personnel to address the surge in patients seeking care. The risk of this situation occurring in other countries is highlighted by the propensity for high infectiousness and asymptomatic spread. To protect patients and the community-at-large, research is urgently needed to guide quarantine and treatment strategies for COVID-19.

Morbidity and mortality from COVID-19 is associated with the development of fulminant respiratory failure. Recent data suggests death rates as high as 38% among those requiring ICU care, many of whom developed Acute Respiratory Distress Syndrome (ARDS). However, it is currently unknown which patients are at risk of severe disease. Diagnostic tools are urgently needed to detect immunologic and physiologic disease responses to identify infection in asymptomatic individuals and to identify infections on the trajectory to ARDS. Furthermore, the infectious reservoirs of SARS CoV-2 remain unclear although children may be important reservoirs given children's relatively mild disease course as well as prolonged viral shedding from both respiratory and stool specimens. This protocol aims to address these critical knowledge gaps and future questions relevant to COVID-19 clinical management.

INPATIENT Enrolled inpatient individuals will have whole blood, 1 RNA tube, serum, nasopharyngeal (NP) or oropharyngeal (OP) swabs collected at enrollment. Subsequent blood (whole blood, serum, or plasma) collections solely for research among hospitalized patients will be a maximum of 10 mL per day. This will generally follow a schedule of day 0/1, 3, 7 and weekly while hospitalized. Subsequent collections after hospital discharge occur at 1 month, 3 months, 6 months, 9 months, and 12 months.

Clinical data from routine clinical care that will be recorded include but are not limited to:

* Symptoms
* Comprehensive medical history
* Medications
* Physical exam including vital signs and oxygen administration
* Clinical and microbiology labs performed during (Complete Blood Count (CBC), chemistries, lactate, blood culture results, HIV results)
* Images and/or imaging results from hospital record

OUTPATIENT After enrollment, a shipping coordinator will contact the participant to confirm participant's willingness to participate and to verify the shipping address to which a study self-testing kit will be mailed. This kit will contain a thermometer, pulse oximeter, gloves, NP and OP swabs (for days 0, 3, 7, 14), 4 viral transport media into which the swabs will be put after testing, Tasso and/or dried blood spot testing kits, Oracol (oral fluid collection tube).

Participants with confirmed or suspected COVID-19, 18 years of age and older will be followed with sample self-collection. Sample self-collection will occur on Day 0, which should occur within 24-48 hours of enrollment. Sample self-collection will also occur on days 3 , 7, 14,(-1/+1) and 28 days (+32). Participants with persistent symptoms will have an additional collection date at 21 days (-2/+2) if feasible. Participants will be advised to do this by themselves and not ask others for assistance. A self-testing kit would include clear instructions for self-collection of samples. This may include respiratory, oral fluid, and dried blood spot/painless capillary blood collection depending on availability of resources. Depending on shipping resources, samples will be temporarily stored in the participant's personal freezer. Vital signs (e.g., heart rate, oxygen saturation, temperature) will be collected by participants with positive COVID-19 results using devices provided by the study when resources are available (e.g. portable pulse oximeter and/or thermometer). Questionnaires for demographic, medical history, socioeconomic, mental health, household contacts, and housing situation will be administered electronically or by study staff depending on the study participant's situation. A standard symptom questionnaire will be administered at every sampling time point either electronically or by study staff including day 28.

ELIGIBILITY:
INPATIENT

Inclusion criteria:

* Newborns to adults 18 years of age or older AND
* Hospitalized with a suspected or proven infection with SARS-CoV-2.

Exclusion criteria:

* Confirmed diagnosis of a pathogen unrelated to the objectives of this study AND no indication or likelihood of co-infection with a relevant pathogen. OR
* Refusal by participant, parent or appropriate representative. OR
* Individuals with any condition or major comorbidity that the study investigators believe will compromise the patient's ability to comply with the requirements of the study.

OUTPATIENT

Inclusion criteria:

* Adults 18 years of age or older AND
* Suspected or proven infection with SARS-CoV-2 pending test results from any Johns Hopkins Health system testing site including individuals who ultimately test negative (for use as negative controls.)

Exclusion criteria:

* Refusal by participant, parent or appropriate representative. OR
* Individuals with any condition or major comorbidity that the study investigators believe will compromise the patient's ability to comply with the requirements of the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: INPATIENT Confirmed and suspected patients with COVID-19 presenting to a Johns Hopkins Health System hospital
  OUTPATIENT Identification of Potential Participants / Recruitment Persons > age 18 who received testing for SARS-CoV-2 after attending a Johns Hopkins Health System Testing site.
Sampling Method: Non-Probability Sample
Enrollment: 702 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Duration of viral shedding | 3 months
  SARS-CoV-2 Reverse transcription polymerase chain reaction (RT-PCR) and viral culture will be performed on prospectively collected samples to determine presence and Ct of viral RNA and presence or absence of cultivable virus in assessing how long virus is shed (in days).

SECONDARY OUTCOMES:
Incidence of comorbidities | 12 months
  Incidence of comorbidities (chronic kidney disease, lung disease, cardiovascular disease, venous thromboembolism) will be determined.
Treatment response as assessed by survival | 1 month
  Survival with the use of treatment with off-label therapeutics or management strategies will be assessed.
Treatment response as assessed by survival | 3 months
  Survival with the use of treatment with off-label therapeutics or management strategies will be assessed.
Mortality of COVID-19 | 12 months
  Survival rates overall will be determined in assessing the mortality of COVID-19.
Change in lung ultrasound score | Baseline and 1 month
  Changes in a lung ultrasound score (LUS) over time will be calculated and evaluated for prediction of disease severity defined by the World Health Organization COVID-19 ordinal scale (clinical status on an ordinal scale from 0 to 8 with higher scores meaning worse outcome).
Change in immunoglobulin M (IgM) antibody levels in serum | Baseline, one month, and every three months up to 12 months
  Change in IgM antibody levels in serum will be determined for description of host response.
Change in immunoglobulin G (IgG) antibody levels in serum | Baseline, one month, and every three months up to 12 months
  Change in IgG antibody levels in serum will be determined for description of host response.
Change in immunoglobulin A (IgA) antibody levels in serum | Baseline, one month, and every three months up to 12 months
  Change in IgA antibody levels in serum will be determined for description of host response.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Sauer, MS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The COVID-19 Biospecimen Committee evaluates requests from researchers for accessing serum or plasma from COVID-19 patients. The committee's default position will be for investigators to receive premade specimen collections for pilot studies with requests for custom made collections considered after pilot studies are completed.
  https://ictr.johnshopkins.edu/coronavirus/biospecimencommittee/